CLINICAL TRIAL: NCT07287891
Title: Lost in the Labyrinth: Predicting Central Neurological Causes of Vertigo Dizziness and Unsteadiness in the Emergency Department. A Multicentre Cross-sectional Observational Study
Acronym: VERTIGO
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Marco Bonzano, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: VERTIGO
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-02

CONDITIONS: ED With Vertigo; Dizziness; Unsteadiness
MeSH Terms: conditions — Dizziness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients presenting at the ED with vertigo, dizziness, and unsteadiness: Patients presenting to the ED with vertigo/ dizziness
  Interventions: Diagnostic Test: Bedside examination of Vertigo

INTERVENTIONS:
Diagnostic Test: Bedside examination of Vertigo — ED visit comprehensive of bedside examination of vertigo performed by trained EP or emergency medicine residents

SUMMARY:
This study will assess the sensitivity and specificity of the bedside examination algorithm performed by ED physicians. Finally, it aims to identify predictors of a central cause of the symptoms. This will consequently reduce the rate of misdiagnosis as well as the costs and length of stay due to inappropriate neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting at the ED with vertigo, dizziness or unsteadiness
* >= 18 years of age
* Patients able to give their consent

Exclusion Criteria:

* Patients with dementia
* Bedridden patients (for causes other than the current symptoms)
* Patients with obvious neurological findings presenting with vertigo but with suspected stroke at triage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at the ED with vertigo, dizziness or unsteadiness
Sampling Method: Non-Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2027-02-26 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
The AUC of the bedside examination algorithm performed by ED physicians | up to 36 months

SECONDARY OUTCOMES:
identification of predictors of true positive patients | up to 36 months
  Predictors of true positive patients can help to stratify patients with vertigo for the risk of stroke.
evaluation of number of neuroimaging tests (TC and angio-TC) performed to patients with vertigo in the ED.tests performed | up to 36 months
  to study the use of ED resources for these patients in terms of number of neuroimaging tests performed.

CONTACTS AND LOCATIONS:
Locations (1):
- SC Pronto Soccorso e Medicina d'Urgenza, Fondazione IRCCS Policlinico San Matteo, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No